CLINICAL TRIAL: NCT04819373
Title: A Phase 2, Open-label, Multi-Arm Trial to Evaluate the Efficacy and Safety of BDB001 in the Treatment of Subjects With Advanced Solid Tumors That Have Progressed on Anti-PD-1 or Anti-PD-L1 mAb Treatment
Brief Title: BDB001-201: A Clinical Study of BDB001 in Patients With PD-(L)1 Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDB001-201
Record Dates: First submitted 2021-01-18; First posted 2021-03-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
Keywords: TLR, Immuno-oncology
MeSH Terms: conditions — Neoplasms | interventions — BDB001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BDB001 (Experimental): BDB001 will be administered intravenously as monotherapy in subjects with histologically-confirmed unresectable or metastatic solid tumors that have progressed on anti-PD-1 or anti-PD-L1 mAb treatment either as monotherapy or in combination with other therapies.
  Interventions: Drug: BDB001

INTERVENTIONS:
Drug: BDB001 — BDB001 is an immunotherapy agent.

SUMMARY:
BDB001-201 is a multi-center, open-label, Phase II clinical trial to evaluate the efficacy and safety of BDB001 in the treatment of subjects with advanced solid tumors that have progressed on anti-PD-1 or anti-PD-L1 mAb treatment.

DETAILED DESCRIPTION:
BDB001-201 is a multi-center, open-label, multi-arm Phase II study evaluating an experimental immunotherapy drug called BDB001. BDB001 is a Toll-like receptor 7/8 (TLR7/8) agonist delivered intravenously to systemically activate the innate and adaptive immunity in the treatment of various tumors.

The objectives of this study are to evaluate the efficacy, safety and tolerability of intravenous BDB001 administered as monotherapy in subjects with histologically-confirmed unresectable or metastatic solid tumors that have progressed on anti-PD-1 or anti-PD-L1 mAb treatment either as monotherapy or in combination with other therapies.

The following tumor types may be included in the trial: Non-Small Cell Lung Cancer (NSCLC); Cutaneous Squamous Cell Carcinoma (cSCC); Head and Neck Squamous Cell Carcinoma (HNSCC); Melanoma; Merkel Cell Carcinoma (MCC); Renal Cell Carcinoma (RCC); Urothelial Carcinoma; other types of solid tumors at the discretion of the Sponsor. Each tumor type will be analyzed independently

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Histologically or cytologically confirmed: Cutaneous SCC, Head and Neck SCC, Melanoma, Merkel Cell Carcinoma, NSCLC, Renal Cell Carcinoma, or Urothelial Carcinoma. Other tumor types will be allowed at Sponsor's discretion.
2. Tumor progression on the most recent line of treatment with anti-PD-1 or anti-PD-L1 mAb as monotherapy or in combination.
3. Eastern Cooperative Oncology Group (ECOG) score of 0 - 2
4. At least 1 lesion with measurable disease at baseline
5. Availability of a lesion for biopsy and consent to allow pre-treatment tumor biopsy.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Greater than 4 lines of prior DNA-damaging chemotherapies.
2. Uncontrolled CNS metastases.
3. Active autoimmune disease.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by Objective Response Rate | Approximately up to 2 years
  Objective Response Rate

SECONDARY OUTCOMES:
Efficacy as measured by Disease Control Rate | Approximately up to 2 years
  Disease Control Rate (DCR)
Efficacy as measured by Progression-Free Survival (PFS) | 3 months through approximately 2 years
  Progression-Free Survival (PFS): The time from first day of study drug infusion to the first documented disease progression or death due to any cause, whichever occurs first.
Evaluate Duration of Response (DoR) | 3 months through approximately 2 years
  Duration of Response (DoR): For subjects who demonstrate CR (Complete Response) or PR (Partial Response) per irRECIST (Immune-related Response Evaluation Criteria In Solid Tumors), DoR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Efficacy as measured by Time-to-Treatment Failure (TTF) | Approximately up to 2 years
  Time-to-Treatment Failure (TTF)
Efficacy as measured by Overall Survival (OS) | Approximately up to 2 years
  Overall Survival (OS)
Efficacy as measured by RECIST 1.1 (ORR, DCR, PFS, and DoR) | 3 months through approximately 2 years
  Evaluate ORR, DCR, PFS, and DoR per RECIST 1.1
Safety and Tolerability of BDB001 | Approximately up to 2 years
  Evaluate Adverse events (AEs) and AEs causing drug discontinuation
Evaluate Biomarkers | Approximately up to 1.5 years
  Evaluate blood samples and tumor biopsy samples for signs of systemic and local immunologic changes by measuring cytokines and transcriptional RNA, and by immunophenotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Raftopoulos, MD, Study Chair — Eikon Therapeutics
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No